CLINICAL TRIAL: NCT00773942
Title: Design & Evaluation of a Medication Therapy Management Program to Improve Patient Safety in Medicare Beneficiaries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Duke University (Other); Baylor Research Institute (Other); RTI International (Other)
Responsible Party: Principal Investigator, Daniel R. Touchette, Professor of Pharmacy, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-0305; HHSA290200500381 T02 (Other Grant/Funding Number: AHRQ)
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Chronic Illness; Adverse Effects; Medication Errors; Elderly Patients
Keywords: Medication therapy management; Pharmacist; Chronic care; Medicare; Medicaid; Medication reconciliation; Adverse drug events; Drug related problems
MeSH Terms: conditions — Chronic Disease; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care (No Intervention): Study subjects receive usual care, without the intervention.
- Basic medication therapy management (Experimental): Subjects in this arm will receive medication reconciliation and drug related problem assessment by a medication therapy management clinician utilizing patient interview alone.
  Interventions: Behavioral: Basic medication therapy management
- Enhanced medication therapy management (Experimental): Subjects in this arm will receive medication reconciliation and drug related problem assessment by a medication therapy management clinician utilizing patient interview and a brief chart synopsis including patient medical history, medication history, and relevant laboratory information.
  Interventions: Behavioral: Enhanced medication therapy management

INTERVENTIONS:
Behavioral: Basic medication therapy management — Subjects in this arm will receive medication reconciliation and drug related problem assessment by a medication therapy management clinician utilizing patient interview alone.
  Arms: Basic medication therapy management
Behavioral: Enhanced medication therapy management — Subjects in this arm will receive medication reconciliation and drug related problem assessment by a medication therapy management clinician utilizing patient interview and chart information.
  Arms: Enhanced medication therapy management

SUMMARY:
The purpose of this study is to determine if a medication therapy management program designed to reconcile a patient's medications and identify and resolve drug related problems can reduce adverse drug events and other measures of safety and improve patient satisfaction.

DETAILED DESCRIPTION:
This study will be a multicenter, prospective, randomized study of usual care (Arm 1; control group) compared with usual care plus medication reconciliation by patient interview and a drug related problem assessment (Arm 2; Basic MTM) and usual care plus medication reconciliation by patient interview with additional information obtained from the patient chart and drug related problem assessment (Arm 3; Enhance MTM). Approximately 600 patients will be enrolled in this study, 200 in each study arm. Two hundred potential subjects will be recruited at each of the three participating sites: the UIC Medical Center, Baylor Health Care System, and Duke Primary Care Research Consortium. For inclusion in the study, patients must be at least 65 years old, primarily uses English for written and oral communication, have 3 or more comorbid conditions from a list of conditions (see table 1 of protocol), have two or more physician office visits at one or more affiliated clinics in the past year, have received 8 or more different chronic prescription medications over the six months prior to the enrollment period, have a telephone line and agree to maintain if for at least 6 months, and have a situation placing him/her at risk for a drug related problem (see protocol for list). Subjects unable to demonstrate comprehension of the informed consent, with a terminal condition, or those enrolled in an MTM program where medication reconciliation and/or assessment of drug related problems has occurred in the previous 12 months will be excluded from enrolling in the study.

Patients in the control group will participate in the baseline study visit, will continue to have access to the regular scheduled physician clinic visit and their prescription filled at the UIC pharmacy, and will participate in the telephone survey after the sixth month of the study. Patients in the Arms 2 and 3 intervention groups will participate in the baseline visit, will be asked to participate in two clinic visits with an MTM clinician, and will be asked to answer two telephone surveys (at 3 months and at 6 months after enrollment).

ELIGIBILITY:
Inclusion Criteria:

* Be at least 65 years old at enrollment
* Primarily uses English language for written and oral communication
* Have three or more comorbid conditions associated with increased healthcare utilization (Diabetes Mellitus, Congestive Heart Failure, Asthma, Hypertension, Dyslipidemia, COPD, Coronary Artery Disease, Chronic Renal Failure, Arthritis, Depression, Dementia, Chronic Pain, Conditions requiring anticoagulation with warfarin)
* Have visited a physician at one or more of the clinics on a regular basis (defined as two or more clinic visits over one year prior to the study start) for these conditions
* Have received 6 or more different chronic prescription medications over the six months prior to the enrollment period
* Have a telephone line and agree to maintain it for at least six months
* Have one of the following situations placing him/her at risk for a DRP (Any ER visit in past 30 days or Urgent Care visit in past 30 days leading to a change in medication or change in medication dose; New physician visit in past 30 days; Hospitalization in past 30 days; Invasive procedure (a procedure requiring substantive changes to medication taking practices or which requires informed consent) in past 30 days; Change in medication in past 30 days; Three or more providers seen in the past year

Exclusion Criteria:

* Terminal condition, where life expectancy is less than 6 months
* Patients already enrolled in an MTM program where medication reconciliation and/or assessment of DRPs has occurred in the previous 12 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 637 (Actual)
Dates: Start 2007-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Adverse Drug Events | 3 and 6 months
  ADEs will be assessed via patient telephone interview using a tool modified from Jarernsiripornkul et al

SECONDARY OUTCOMES:
Emergency department visits | 6 months
  The number of ED visits collected by a blinded study investigator 180 days via patient self report obtained during a telephone interview
Hospitalizations | 6 months
  The number of hospitalizations collected by a blinded study investigator 180 days via patient self report obtained during a telephone interview
Drug related problems | 3 and 6 months
  The number and types of DRPs will be collected from form completed by MTM clinician
Discrepancies in medication list, intervention arms compared with best possible medication history | 6 months
  Differences observed in MTM intervention medication list and a "Best Possible Medication History," as developed by a formal process and conducted by a study investigator.
Patient satisfaction with care. | 6 months
  Patient self-reported satisfaction with care, obtained using the Pharmacutical Care Questionnaire administered via telephone interview. Overall satisfaction of care assessed using a 3-item questionnaire administered during telephone interview.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Touchette, PharmD, MA, Principal Investigator — University of Illinois at Chicago
Locations (3):
- United States (3):
  - University of Illinois at Chicago, Chicago, Illinois
  - Duke University Health System, Durham, North Carolina
  - Baylor Health Care System, Dallas, Texas

REFERENCES:
- [Background] Masica AL, Touchette DR, Dolor RJ, Schumock GT, Kliethermes MA, Rodgers PT, Craft JL, Choi YK, Lux LJ, Smith SR. Evaluation of a Medication Therapy Management Program in Medicare Beneficiaries at High Risk of Adverse Drug Events: Study Methods. In: Henriksen K, Battles JB, Keyes MA, Grady ML, editors. Advances in Patient Safety: New Directions and Alternative Approaches (Vol. 4: Technology and Medication Safety). Rockville (MD): Agency for Healthcare Research and Quality (US); 2008 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK43763/ PMID 21249958
- [Derived] Touchette DR, Masica AL, Dolor RJ, Schumock GT, Choi YK, Kim Y, Smith SR. Safety-focused medication therapy management: a randomized controlled trial. J Am Pharm Assoc (2003). 2012 Sep-Oct;52(5):603-12. doi: 10.1331/JAPhA.2012.12036. PMID 23023840
- [Derived] Dolor RJ, Masica AL, Touchette DR, Smith SR, Schumock GT. Patient safety-focused medication therapy management: challenges affecting future implementation. Am J Manag Care. 2012 Jul 1;18(7):e238-44. PMID 22823552